CLINICAL TRIAL: NCT05081206
Title: Comparison of the Manually Controlled Propofol Infusion and Target Controlled Infusion Anesthesia for One Day Surgery in Pediatric Patients
Brief Title: Comparison of the Manually Controlled Propofol Infusion and Target Controlled Infusion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital (Other)
Responsible Party: Principal Investigator, Irina Milojevic, Chief of the Anesthesiology and Reanimatology Department, University Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TirsovaChildrensH
Record Dates: First submitted 2021-08-10; First posted 2021-10-18 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Propofol Anesthesia in Children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manually controlled (Experimental)
  Interventions: Drug: Propofol infusion via manually controlled pump.
- Target controlled (Experimental)
  Interventions: Drug: Propofol infusion via target controlled pump.

INTERVENTIONS:
Drug: Propofol infusion via manually controlled pump. — Patients will receive propofol bolus 2.5-3 mg/kg, for anesthesia induction and anesthesia maintenance was continued according to the Mc Farlan scheme, meaning continuous propofol infusion is used, with gradual reduction of the infusion speed in timely manner, depending on the duration of surgery: 15mg/kg/h...13mg/kg/h...11mg/kg/h...9mg/kg/h...6mg/kg/h.
  Arms: Manually controlled
Drug: Propofol infusion via target controlled pump. — Pedfusor model was used for delivering target controlled plasma concentration, with target concentration for anesthesia induction of 4 mcg/kg body weight and then 3 mcg/kg.
  Arms: Target controlled

SUMMARY:
Patients 1 to 8 years of age, American Society of Anesthesiologist score 1 and 2, planned for elective, one day surgery: inguinal hernia repair, hydrocele surgery, testis retention surgery, varicocele and phimosis surgery, and parents or legal guardians will be asked to sign written informed consent for participation in the study. Exclusion criteria will be: confirmed propofol allergies, mitochondrial disease, disease of lipid and carbohydrate metabolism, neurological disorders, treated psychiatric comorbidities, hypertension.

All participants will be randomly assigned to two groups: one in which manually controlled propofol infusion will be used (MC group) and the other with target controlled infusion (TC group). After anesthesia induction depth of anesthesia during surgery will be measured using bispectral index (BIS), continuously. As a part of routine monitoring noninvasive blood pressure monitoring will be measured, and recorded in three time points, as well as heart rate. Time will be measured from the moment when propofol infusion was stopped till tracheal extubating.

DETAILED DESCRIPTION:
Prospective, randomized controlled study will be done at the University Children's Clinic. For the study ethical board approval was requested. Pediatric patients, planned for elective, one day surgery, requiring intubation with signed informed consent will be randomly assigned to two groups First in which manually controlled propofol infusion will be used (MC group) and the other with target controlled infusion (TC group).

All participants will be premedicated half an hour before anesthesia induction with midazolam orally in dose of 0.5mg/kg body weight. Intravenous cannula will be placed 20-30 minutes later, and participants will receive atropine in dose of 0,02mg/kg intravenously, and fentanyl 1mcg/kg intravenously. In the MC group participants will receive propofol bolus 2.5-3 mg/kg, for anesthesia induction and anesthesia maintenance will be done according to the Mc Farlan scheme. In TC group Pedfusor model will be used, with target concentration for anesthesia induction of 4 mcg/kg body weight and anesthesia maintenance of 3 mcg/kg. In all participants remifentanil in dose of 0.4mcg/kg/min will be used as analgesic, and cisatracurium 0.15mg/kg was muscle relaxant, for anesthesia induction. At the end of surgery, before remifentanil infusion is stopped, all patients will receive 0.5 mg/kg of ketorolac. If BIS values are out of the40-60 range during anesthesia, in MC group infusion rate will be changed and in TC group set plasma concentration (Cp) will be corrected. In case of heart rate increase or decrease for more than 20% compared to initial values, speed of remifentanil infusion will be decreased or increased, respectively. All participants will have standard monitoring during anesthesia: percutaneous saturation, end tidal concentration of carbon dioxide measurement, three channel electrocardiography, noninvasive blood pressure monitoring, and continuous BIS measurement. Propofol infusion will be stopped 5 minutes before expected end of surgery, and remifentanil infusion will be stopped at the end of surgery. Time will be measured from the moment when propofol infusion was stopped till tracheal extubating.

ELIGIBILITY:
Inclusion Criteria:

* ASA score 1 and 2.
* Planned for elective, one day surgery: inguinal hernia repair, hydrocele surgery, testis retention surgery, varicocele and phimosis surgery,
* Signed written informed consent for participation in the study by parent and/or legal guardian.

Exclusion Criteria:

* Confirmed propofol allergies.
* Mitochondrial disease
* Disease of lipid and carbohydrate metabolism
* Neurological disorders
* Treated psychiatric comorbidities
* Hypertension.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Depth of anesthesia comparison between two experimental groups. | From anesthesia induction till extubation, every minute up to 90 minutes.
  Depth of anesthesia will be measured with continuous bispectral index and compared between two experimental groups.

SECONDARY OUTCOMES:
Comparison of blood pressure between two experimental groups. | At 0 and 20 minutes during anesthesia and 5 minutes after discontinuation of propofol infusion.
  Blood pressure will be measured in three specified time points during anesthesia, and the values will be compared between two experimental groups.
Comparison of heart rate between two experimental groups. | At 0 and 20 minutes during anesthesia and 5 minutes after discontinuation of propofol infusion.
  Heart rate will be measured in three specified time points during anesthesia, and the values will be compared between two experimental groups.
Time to tracheal extubation comparison between two experimental groups. | 5 to 15 minutes after discontinuation of propofol infusion
  Time to tracheal extubation will be measured after propofol infusion termination in both experimental groups and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No